CLINICAL TRIAL: NCT07173634
Title: Comparison of Speaking Valve Trial Versus Capping Trial in the Decannulation Process for Patients With Prolonged Disorders of Consciousness: A Randomized Controlled Study
Brief Title: Speaking Valve Trial vs. Capping Trial for Tracheostomy Decannulation in Prolonged Disorders of Consciousness
Acronym: SPEAK-CAP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hongying Jiang (Other)
Collaborators: Beijing Rehabilitation Hospital (Other); Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor-Investigator, Hongying Jiang, Principal Investigator, Capital Medical University
Organization: Capital Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-hxkf-s&tc
Record Dates: First submitted 2025-09-04; First posted 2025-09-15 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Prolonged Disorders of Consciousness
Keywords: Prolonged disorders of consciousness; Decannulation; Speaking wave; Capping; Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Speaking Valve (SV) Group (Experimental): Stepwise speaking valve tolerance: 0.5h → 1h → 2h → 4h. Decannulation if: Tolerates a 4-hour speaking valve trial with pulse oxygen saturation (SpO₂) ≥ 95%, breathing rate (RR) < 20/min, and no signs of distress during the 4-hour trial.
  Interventions: Other: Speaking Valve Trial
- Capping Group (Active Comparator): Gradual capping: 1 hour → 4 hours → 6 hours → 12 hours → 24 hours → 48 hours. Decannulation if: Tolerates 48 hours of capping with SpO₂ ≥95%, respiratory rate (RR) <20/min, and no distress during the 48-hour trial.
  Interventions: Other: Capping Trial

INTERVENTIONS:
Other: Speaking Valve Trial — The speaking valve group ascertains a patient's eligibility for decannulation following the results of the speaking valve test. A patient who can endure a 4-hour trial with a speaking valve, maintaining a pulse oxygen saturation (SpO₂) of at least 95%, a breathing rate (RR) below 20 per minute, and exhibiting no signs of distress throughout the trial, qualifies for decannulation.
  Arms: Speaking Valve (SV) Group
Other: Capping Trial — The capping valve group determines a patient's eligibility for decannulation based on the results of the capping test. A patient who can tolerate 48 hours of capping with a pulse oxygen saturation (SpO₂) of ≥95%, a breathing rate (RR) of <20/min, and no signs of distress during the 48-hour trial, is eligible for decannulation.
  Arms: Capping Group

SUMMARY:
To assess whether the speaking valve trial, when employed as an indicator for extubation during the removal of tracheostomy tubes in patients with chronic consciousness disorder, provides superior benefits and heightened sensitivity relative to the conventional capping trial, thereby enhancing the overall extubation process.

DETAILED DESCRIPTION:
Patients with chronic consciousness disorder who require long-term mechanical ventilation and airway protection commonly undergo tracheostomy. However, tracheostomy tubes can cause inflammation, stenosis, excessive coughing, and swallowing dysfunction. Removing the tracheostomy tube, or extubation, can prevent long-term complications such as tracheal stenosis, tracheomalacia, vocal cord injury, and accidental extubation. Additionally, it enhances patient comfort, appearance, swallowing function, communication ability, and social integration. Therefore, for clinically stable patients with chronic consciousness disorder who can breathe spontaneously, have effective cough reflexes, and are capable of protecting their airways, early tube removal is advisable.In current extubation protocols, the capping trial is predominantly used to assess whether patients can tolerate tracheostomy tube removal. There have also been reports of studies using speaking valves as an alternative to the capping trial, but no direct comparison has been made between the two methods. Patients who can tolerate capping for 24 hours are generally considered suitable for tracheostomy tube removal. A speaking valve is a one-way valve placed at the end of the tracheostomy tube that directs airflow to the upper airway when the cuff is deflated. Studies have found that patients undergoing speaking valve training benefit in terms of vital signs, airway secretions, sense of smell, weaning from mechanical ventilation, post-tracheostomy extubation, hospital stay duration, and quality of life. However, it remains unclear whether this method can improve the success rate of extubation assessment in patients with chronic consciousness disorder. This study compares speaking valve training and the traditional capping trial in post-tracheostomy patients with chronic consciousness disorder, evaluating differences in extubation tolerance, extubation success rate, time to extubation, hospital stay duration, and improvement in consciousness levels.

Parazacco spilurus subsp. spilurus

ELIGIBILITY:
Inclusion Criteria:

1. Adults (18-80 years) with tracheostomy
2. Prolonged DoC (>28 days) confirmed by CRS-R score >0
3. Ventilator-free >48h
4. PaCO₂ <60 mmHg
5. PCF ≥100 L/min
6. No sepsis/organ failure
7. Controlled pulmonary infection
8. Written informed consent by legal representative

Exclusion Criteria:

1. Intolerance to cuff deflation:
2. SpO₂ <93% on O₂ supplementation OR Respiratory rate >20/min for >5min
3. Severe tracheal stenosis (>50% lumen occlusion on CT)
4. Death within 2 weeks post-enrollment
5. Participation in conflicting interventional trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Decannulation rate | At decannulation
  Proportion passing full protocol
Decannulation success rate | At 48 h post decannulation
  (Decannulation - Decannulation failure ) / Decannulation

SECONDARY OUTCOMES:
Time to decannulation | 1year
  Days from randomization to successful tube removal
Hospital stay duration | Up to 6 months
  Days from randomization to discharge without tracheostomy care
CRS-R change rate | 3 months
  (Post-decannulation score - Baseline)/Baseline
Airway safety score1 | 48h post-decannulation
  Pulse oxygen saturation (SpO₂) fluctuation, minimum value0%, maximum value 100%, the larger the value, the better the result
Airway safety score 2 | 48h post-decannulation
  Blood carbon dioxide partial pressure (pCO₂) , normal range 35-45mmHg. Within the normal range it is good, the greater the deviation from the normal range, the worse the result the larger the value, the better the result.

CONTACTS AND LOCATIONS:
Overall Officials: Hongying Jiang, Study Chair — Beijing Rehabilitation Hospital, Capital Medical University, Beijing

IPD SHARING:
Plan to Share IPD: No